CLINICAL TRIAL: NCT00614744
Title: Evaluation of Systemic Hypothermia Initiated After 6 Hours of Age in Infants ≥36 Weeks Gestation With Hypoxic-Ischemic Encephalopathy: A Bayesian Evaluation. A Protocol for the NICHD Neonatal Research Network
Brief Title: Late Hypothermia for Hypoxic-Ischemic Encephalopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NICHD-NRN-0038; U10HD036790 (NIH); U10HD021364 (NIH); U10HD021373 (NIH); U10HD021385 (NIH); U10HD027851 (NIH); U10HD027853 (NIH); U10HD027856 (NIH); U10HD027871 (NIH); U10HD027880 (NIH); U10HD027904 (NIH); U10HD034216 (NIH); U10HD040492 (NIH); U10HD040689 (NIH); U10HD053089 (NIH); U10HD053109 (NIH); U10HD053119 (NIH); U10HD053124 (NIH); UL1RR024139 (NIH); UL1RR025744 (NIH); UL1RR024979 (NIH); U10HD068244 (NIH); 1U10HD068263-01 (NIH); U10HD068270 (NIH); U10HD068278 (NIH); U10HD068284 (NIH)
Record Dates: First submitted 2008-02-11; First posted 2008-02-13 (Estimated); Results first posted 2017-08-07 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-02

CONDITIONS: Infant, Newborn; Hypoxia, Brain; Hypoxia-Ischemia, Brain; Encephalopathy, Hypoxic-Ischemic; Hypoxic-Ischemic Encephalopathy; Ischemic-Hypoxic Encephalopathy
Keywords: NICHD Neonatal Research Network; Hypoxic-ischemic encephalopathy (HIE); Hypothermia; Neonatal depression; Perinatal asphyxia
MeSH Terms: conditions — Hypoxia, Brain; Hypoxia-Ischemia, Brain; Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Whole-body Hypothermia (Experimental): Induced Whole-body hypothermia (with a target esophageal temperature of 33.5°C) for 96 hours
  Interventions: Procedure: Hypothermia
- Normothermia (Active Comparator): Normothermic Control group (with esophageal temperature at or near 37.0°C) for 96 hours
  Interventions: Procedure: Normothermic Control

INTERVENTIONS:
Procedure: Hypothermia — Induced Whole-body hypothermia (with a target esophageal temperature of 33.5°C) for 96 hours
  Arms: Whole-body Hypothermia
Procedure: Normothermic Control — Normothermic Control group (with esophageal temperature at or near 37.0°C) for 96 hours
  Arms: Normothermia

SUMMARY:
This study is a randomized, placebo-controlled, clinical trial to evaluate whether induced whole-body hypothermia initiated between 6-24 hours of age and continued for 96 hours in infants ≥ 36 weeks gestational age with hypoxic-ischemic encephalopathy will reduce the incidence of death or disability at 18-22 months of age. The study will enroll 168 infants with signs of hypoxic-ischemic encephalopathy at 16 NICHD Neonatal Research Network sites, and randomly assign them to either receive hypothermia or participate in a non-cooled control group.

DETAILED DESCRIPTION:
Hypoxic-ischemic encephalopathy (HIE) is a rare, but life-threatening condition characterized by acute or subacute brain injury due to asphyxia. In most cases the underlying cause and timing of injury are unknown, but many cases are diagnosed at or shortly after birth.

According to the World Health Organization, more than 722,000 children died from birth asphyxia and birth trauma worldwide in 2004. An estimated 50-75 percent of infants with severe (stage 3) HIE will die, with 55 percent of these deaths occurring in the first month.

The incidence of long-term complications depends on the severity of HIE. Up to 80 percent of infants who survive stage 3 HIE develop significant long-term neurological disabilities - mental retardation, epilepsy, and cerebral palsy with hemiplegia, paraplegia, or quadriplegia; 10-20 percent develop moderately serious disabilities; and up to 10 percent are normal.

Because animal data suggests that brain injury from HIE evolves over several hours to days after the initial asphyxic insult, induced hypothermia holds promise as a neuroprotective therapy. Additional trials are needed to help define the most effective cooling strategies.

With this in mind, and knowing that many babies with HIE arrive at neonatal intensive care units several hours after birth, this study will evaluate the safety and efficacy of initiating hypothermia 6-24 hours after birth.

Study subjects: Infants born at 36 0/7ths weeks or greater gestational age that have been diagnosed with neonatal depression, perinatal asphyxia, or encephalopathy. The goal is to enroll 168 subjects.

Stratification: After informed consent is obtained, infants will be randomized to either a hypothermia arm (with a target esophageal temperature of 33.5°C) or a control arm (37.0°C) for 96 hours. Enrolled infants will be stratified by age of enrollment (≤ 12 and > 12 hours) and stage of encephalopathy (moderate or severe).

Informed Consent: Parents of eligible infants will be approached for consent to enroll in the study if the infant has a high probability of acute hemodynamic compromise, as defined above. Subsequent screening will determine whether the infant meets all inclusion criteria.

Randomization: eligible and consented infants will be randomly assigned to either a hypothermia intervention group, or a non-cooled (control) group.

Study Intervention: Induced whole-body hypothermia (with a target esophageal temperature of 33.5°C) or a control group (37.0°C) for 96 hours.

Interim Study Interruptions: None to date.

Secondary Study includes determining an association between MRI detectable injury and neurodevelopment at 18-22 months.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at 36 0/7ths weeks gestational age or greater (by best obstetrical estimate)
* Postnatal age between 6 and 24 hours following birth
* Infants with a high probability of acute hemodynamic compromise, such as those with:

  * An acute perinatal event (abruptio placenta, cord prolapse, severe FHR abnormality)
  * An Apgar score ≤ 5 at 10 minutes
  * Continued need for ventilation initiated at birth for at least 10 minutes
  * Cord pH or first postnatal blood gas pH at ≤ 1 hour of ≤ 7.0
  * Base deficit on cord gas or first postnatal blood gas at ≤ 1 hour of ≥ 16 mEq/L
* Infants matching the above criteria who also have an abnormal neurological exam showing the presence of moderate or severe encephalopathy
* Infants whose parents/legal guardians have provided consent for enrollment.

NOTE: These inclusion criteria are identical to the NICHD Neonatal Research Network's 2005 Hypothermia study (see links below), except for the time of entry (6-24 hours vs. < 6 hours of age).

Exclusion Criteria:

* Any infant with a core body temperature (axilla, rectal) less than 34.0°C for greater than 1 hour
* Presence of a known anomaly or chromosomal aberration
* Birth weight < 1,800 grams
* Infant in extremis
* Infants whose parents/legal guardians or attending physician refuse consent

Ages: 6 Hours to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 168 (Actual)
Dates: Start 2008-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abbot R. Laptook, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; Michele C. Walsh, MD MS, Principal Investigator — Case Western Reserve University, Rainbow Babies and Children's Hospital; Ronald N. Goldberg, MD, Principal Investigator — Duke University; Barbara J. Stoll, MD, Principal Investigator — Emory University; Brenda B. Poindexter, MD MS, Principal Investigator — Indiana University; Abhik Das, PhD, Principal Investigator — RTI International; Krisa P. Van Meurs, MD, Principal Investigator — Stanford University; Ivan D. Frantz III, MD, Principal Investigator — Tufts Medical Center; Kurt Schibler, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Waldemar A. Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Edward F. Bell, MD, Principal Investigator — University of Iowa; Kristi L. Watterberg, MD, Principal Investigator — University of New Mexico; Myra Wyckoff, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; Kathleen A. Kennedy, MD MPH, Principal Investigator — The University of Texas Health Science Center, Houston; Roger G. Faix, MD, Principal Investigator — University of Utah; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Richard A. Ehrenkranz, MD, Principal Investigator — Yale University; William Truog, MD, Principal Investigator — Children's Mercy Hospital Kansas City; Barbara Schmidt, MD, MSc, Principal Investigator — University of Pennsylvania; Carl D'Angio, MD, Principal Investigator — University of Rochester; Uday Devaskar, MD, Principal Investigator — University of California, Los Angeles; Pablo Sanchez, M.D, Principal Investigator — Ohio State University
Locations (22):
- United States (22):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California - Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Tufts Medical Center, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - Univeristy of Pennsylvania, Philadelphia, Pennsylvania
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Bonifacio SL, Chalak LF, Van Meurs KP, Laptook AR, Shankaran S. Neuroprotection for hypoxic-ischemic encephalopathy: Contributions from the neonatal research network. Semin Perinatol. 2022 Nov;46(7):151639. doi: 10.1016/j.semperi.2022.151639. Epub 2022 Jun 10. PMID 35835616
- [Derived] Laptook AR, Shankaran S, Barnes P, Rollins N, Do BT, Parikh NA, Hamrick S, Hintz SR, Tyson JE, Bell EF, Ambalavanan N, Goldberg RN, Pappas A, Huitema C, Pedroza C, Chaudhary AS, Hensman AM, Das A, Wyckoff M, Khan A, Walsh MC, Watterberg KL, Faix R, Truog W, Guillet R, Sokol GM, Poindexter BB, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Limitations of Conventional Magnetic Resonance Imaging as a Predictor of Death or Disability Following Neonatal Hypoxic-Ischemic Encephalopathy in the Late Hypothermia Trial. J Pediatr. 2021 Mar;230:106-111.e6. doi: 10.1016/j.jpeds.2020.11.015. Epub 2020 Nov 13. PMID 33189747
- [Derived] Laptook AR, Shankaran S, Tyson JE, Munoz B, Bell EF, Goldberg RN, Parikh NA, Ambalavanan N, Pedroza C, Pappas A, Das A, Chaudhary AS, Ehrenkranz RA, Hensman AM, Van Meurs KP, Chalak LF, Khan AM, Hamrick SEG, Sokol GM, Walsh MC, Poindexter BB, Faix RG, Watterberg KL, Frantz ID 3rd, Guillet R, Devaskar U, Truog WE, Chock VY, Wyckoff MH, McGowan EC, Carlton DP, Harmon HM, Brumbaugh JE, Cotten CM, Sanchez PJ, Hibbs AM, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Effect of Therapeutic Hypothermia Initiated After 6 Hours of Age on Death or Disability Among Newborns With Hypoxic-Ischemic Encephalopathy: A Randomized Clinical Trial. JAMA. 2017 Oct 24;318(16):1550-1560. doi: 10.1001/jama.2017.14972. PMID 29067428
- See also: NICHD Neonatal Research Network — https://neonatal.rti.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multicenter randomized trial to evaluate whether induced hypothermia with body cooling initiated between 6-24 hours of age and continued for 96 hours in infants >= 36 weeks gestation with hypoxic-ischemic encephalopathy will reduce the incidence of death or disability at 18 months of age. Eligible infants were enrolled from 05/06/08 to 07/12/14.
Period: Overall Study
Arm/Group | Whole-body Hypothermia | Normothermia
Started | 83 | 85
Completed | 78 | 79
Not Completed | 5 | 6
Not completed — Lost to Follow-up | 5 | 4
Not completed — Incomplete for Behavior Issues | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Whole-body Hypothermia | Normothermia | Total
Number analyzed (Participants) | 83 | 85 | 168
Age, Customized [Count of Participants; unit: Participants] — Age at Randomization
  Participants
    <= 12 Hours | 26 | 28 | 54
    > 12 Hours | 57 | 57 | 114
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 55 | 102
  Male | 36 | 30 | 66
Level of Encephalopathy [Count of Participants; unit: Participants]
  Moderate | 73 | 78 | 151
  Severe | 10 | 7 | 17
Birthweight [Mean (Standard Deviation); unit: grams] | 3379 (528) | 3303 (553) | 3340 (541)
Length [Mean (Standard Deviation); unit: centimeters] | 51 (3) | 51 (3) | 51 (3)
Gestational Age [Mean (Standard Deviation); unit: weeks] | 39 (2) | 39 (1) | 39 (1)

OUTCOME MEASURES:

1. Primary Outcome: Death or Moderate or Severe Disability
Description: Severe disability was defined by any of the following: a Bayley III cognitive score < 70 or Gross Motor Functional (GMF) Level of 3-5 blindness or profound hearing loss requiring amplification but still unable to follow commands/communicate. Moderate disability was defined as a Bayley III cognitive score between 70-84 and either a GMF level of 2 or a seizure disorder or a hearing deficit.
Time Frame: Birth to 18-22 months corrected gestational age
Population: Does not include 9 lost to follow up and 2 infants without outcome for behavior issues
Measure: Count of Participants; unit: Participants
Arm/Group | Whole-body Hypothermia | Normothermia
Number analyzed (Participants) | 78 | 79
Participants | 19 | 22
Statistical Analysis 1: Comparison: Whole-body Hypothermia vs Normothermia; Whole-body Hypothermia vs. Normothermia (Normothermia is the comparison group); Test type: Superiority — This trial estimated the probability that the intervention has no effect on the outcome (or conversely, the probability that it does), given the data obtained in the trial and any prior evidence; Bayesian log binomial models; Bayesian log binomial models were used to analyze the primary outcome of death or moderate/severe disability; Risk Ratio (RR) = 0.86, 95% CI 2-sided [0.59 to 1.29] — In log binomial models used Normal (0, sd=0.35) neutral prior in the log RR scale. Estimation used Normal weakly informative priors. Reported posterior medians & 95% credible intervals for the RR above instead of confidence intervals; We fitted all Bayesian models via Markov chain Monte Carlo methods (MCMC) using JAGS (version 3.4) and OpenBUGS (3.2.3) in R (version 3.2.5). For each analysis we ran 3 MCMC chains with starting values randomly drawn from the estimated parameters from a frequentist log binomial model. A burn-in of 1,000 iterations was used, with sampling from a further 10,000 iterations for each chain. To monitor convergence, trace plots and the Gelman-Rubin convergence diagnostic (Rhat) were used for all parameters. For all analyses, the trace plots show good mixing of the 3 chains with Rhat < 1.01 for all parameters, indicating convergence

2. Secondary Outcome: Number of Deaths in the NICU and Following Discharge
Time Frame: Birth to 18-22 months corrected gestational age
Population: Does not include 9 lost to follow up and 2 infants without outcome for behavior issues
Measure: Count of Participants; unit: Participants
Arm/Group | Whole-body Hypothermia | Normothermia
Number analyzed (Participants) | 78 | 79
Participants | 9 | 9

3. Secondary Outcome: Number of Infants With Moderate and Severe Disability
Description: Moderate disability will be defined as a Bayley III cognitive score between 70-84 and either a GMF level of 2 or a seizure disorder or a hearing deficit. Severe disability will be defined by any of the following: a Bayley III cognitive score < 70 or Gross Motor Functional (GMF) Level of 3-5 or blindness or profound hearing loss requiring amplification but still unable to follow commands/communicate.
Time Frame: Birth to 18-22 months corrected gestational age
Population: Does not include 9 lost to follow up and 2 infants without outcome for behavior issues
Measure: Count of Participants; unit: Participants
Arm/Group | Whole-body Hypothermia | Normothermia
Number analyzed (Participants) | 78 | 79
Participants | 10 | 13

4. Secondary Outcome: Number of Infants With Mild, Moderate and Severe Disability
Description: Mild disability will be defined by either a Bayley III cognitive score of 70-84 alone or a Bayley III cognitive score >= 85 and any of the following: presence of a GMF level 1 or 2 OR seizure disorder or hearing loss. Moderate disability was defined as a Bayley III cognitive score between 70-84 and either a GMF level of 2 or a seizure disorder or a hearing deficit. Severe disability will be defined by any of the following: a Bayley III cognitive score < 70 OR Gross Motor Functional (GMF) Level of 3-5 OR blindness or profound hearing loss requiring amplification but still unable to follow commands/communicate.
Time Frame: Birth to 18-22 months corrected gestational age
Population: Does not include 9 lost to follow up and 2 infants without outcome for behavior issues
Measure: Count of Participants; unit: Participants
Arm/Group | Whole-body Hypothermia | Normothermia
Number analyzed (Participants) | 78 | 79
Participants | 26 | 25

5. Secondary Outcome: Number of Infants With Any Disability Based on Level of Encephalopathy at Randomization
Description: Mild disability will be defined by either a Bayley III cognitive score of 70-84 alone or a Bayley III cognitive score >= 85 and any of the following: presence of a GMF level 1 or 2OR seizure disorder or hearing loss. Moderate disability was defined as a Bayley III cognitive score between 70-84 and either a GMF level of 2 or a seizure disorder or a hearing deficit. Severe disability will be defined by any of the following: a Bayley III cognitive score < 70 OR Gross Motor Functional (GMF) Level of 3-5 OR blindness or profound hearing loss requiring amplification but still unable to follow commands/communicate.
Time Frame: Birth to 18-22 months corrected gestational age
Measure: Count of Participants; unit: Participants
Arm/Group | Whole-body Hypothermia | Normothermia
Number analyzed (Participants) | 69 | 70
Participants
  Moderate encephalopathy | 24 | 25
  Severe encephalopathy | 2 | 0
  Total | 26 | 25

6. Secondary Outcome: Number of Infants With Non-CNS Organ System Dysfunction
Description: Based on observing presence of organ dysfunction on at least one of the following: Pulmonary (Meconium aspiration syndrome, PPHN, Pulmonary hemorrhage, Pneumonia, Chronic lung disease, ECMO, INO), Cardiovascular (Cardiomegaly, Cardiac failure, Cardiac dysfunction (by echo), Cardiac ischemia (by EKG and/or increased enzymes), Hypotension, Arrhythmia), Renal (Oliguria, Anuria, Dialysis), Gastrointestinal (NEC, Hepatic dysfunction), Hematologic (DIC) and Metabolic (Hypoglycemia, Hypocalcemia, Hypomagnesemia)
Time Frame: Birth to 18-22 months corrected gestational age
Measure: Count of Participants; unit: Participants
Arm/Group | Whole-body Hypothermia | Normothermia
Number analyzed (Participants) | 83 | 85
Participants | 63 | 59

7. Secondary Outcome: Number of Infants With a DNR Order
Time Frame: Birth to 18-22 months corrected gestational age
Measure: Count of Participants; unit: Participants
Arm/Group | Whole-body Hypothermia | Normothermia
Number analyzed (Participants) | 83 | 85
Participants | 7 | 8

8. Secondary Outcome: Number of Infants With a DNR Order and Support is Withdrawn
Time Frame: Birth to 18-22 months corrected gestational age
Measure: Count of Participants; unit: Participants
Arm/Group | Whole-body Hypothermia | Normothermia
Number analyzed (Participants) | 83 | 85
Participants | 6 | 8

9. Secondary Outcome: Number of Infants With a DNR Order That Died
Time Frame: Birth to 18-22 months corrected gestational age
Population: Only infants with DNR order
Measure: Count of Participants; unit: Participants
Arm/Group | Whole-body Hypothermia | Normothermia
Number analyzed (Participants) | 83 | 85
Participants | 5 | 7

10. Secondary Outcome: Number of Infants With Neonatal Seizures, With and Without EEG Abnormalities
Time Frame: Birth to 18-22 months corrected gestational age
Measure: Count of Participants; unit: Participants
Arm/Group | Whole-body Hypothermia | Normothermia
Number analyzed (Participants) | 83 | 85
Participants | 63 | 56

ADVERSE EVENTS:
Time Frame: During study intervention period: 124 hours from baseline (time of insertion of esophageal probe).
Arm/Group | Whole-body Hypothermia | Normothermia
All-Cause Mortality (participants affected / at risk) | 6/83 | 5/85
Serious Adverse Events (participants affected / at risk) | 5/83 | 1/85
Other Adverse Events (participants affected / at risk) | 0/83 | 0/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Whole-body Hypothermia (N=83) | Normothermia (N=85)
Bleeding (Vascular disorders) | 4 (4) | 1 (1)
Alteration of skin integrity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PPHN/Acidosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators must adhere to the Neonatal Research Network Publication policies.